CLINICAL TRIAL: NCT05030649
Title: The Usefulness of Smart-glasses During the Ultrasound-guided Radial Arterial Catheterization in Pediatric Patients by Less Experienced Trainees: a Randomized Controlled Trial
Brief Title: Smart-glasses During the Ultrasound-guided Radial Arterial Catheterization in Pediatric Patients by Trainees
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Principal Investigator, Jin-Tae Kim, Professor, Seoul National University Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Smart Glass A-line Less Exp
Record Dates: First submitted 2021-08-30; First posted 2021-09-01 (Actual); Last update posted 2023-03-07 (Actual); Status verified 2023-03

CONDITIONS: Arterial Line
Keywords: Radial Artery; Vascular Catheters; Smart Glassess; Less experienced
MeSH Terms: interventions — Smart Glasses

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Smart Glasses (Experimental): The real-time ultrasound image is displayed through head-mounted display Moverio BT-300 (Epson Inc., USA) during the radial arterial cannulation.
  Interventions: Device: Smart glasses
- Control (Active Comparator): The real-time ultrasound image is displayed by the ultrasound machine's monitor during the radial arterial cannulation.
  Interventions: Device: Control

INTERVENTIONS:
Device: Smart glasses — The real-time ultrasound image is displayed through head-mounted display Moverio BT-300 (Epson Inc., USA) during the radial arterial cannulation.
  Arms: Smart Glasses
Device: Control — The real-time ultrasound image is displayed by the ultrasound machine's monitor during the radial arterial cannulation.
  Arms: Control

SUMMARY:
The primary objective of the study is to evaluate the effect of smart glasses (Head-mounted display Moverio BT-300 (Epson Inc., USA)) on the first-attempt success rate of radial artery cannulation in pediatric patients by less experienced trainees. This study hypothesizes that the use of smart glasses improves the hand-eye coordination and the first-attempt success rate of radial artery cannulation. This is a single-center, randomized, placebo-controlled study comparing the real-time ultrasound image through smart glasses (intervention group) or the ultrasound machine's monitor (control group) during the radial arterial cannulation in pediatric patients undergoing general anesthesia by less experienced trainees.

ELIGIBILITY:
Inclusion Criteria:

* General anesthesia
* Arterial cannulation for hemodynamic monitoring, multiple blood sample

Exclusion Criteria:

* Unstable vital signs, significant arrhythmia or hypotension, Shock
* High risk of peripheral ischemia
* Skin disease, infection, hematoma, recent cannulation at theradial artery

Max Age: 7 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 122 (Actual)
Dates: Start 2021-09-17 (Actual); Primary Completion 2023-02-07 (Actual); Study Completion 2023-02-07 (Actual)

PRIMARY OUTCOMES:
First attempt success rate | During radial artery cannulation (up to 1 hour)
  Success at the first skin puncture

SECONDARY OUTCOMES:
Size of radial artery | During radial artery cannulation (up to 1 hour)
  Internal diameter of radial artery
depth of radial artery | During radial artery cannulation (up to 1 hour)
  depth of radial artery from the skin
Overall attempt | During radial artery cannulation (up to 1 hour)
  Number of attempt of radial artery cannulation
Ultrasound image time | During radial artery cannulation (up to 1 hour)
  From ultrasound probe application, to get radial artery image on the ultrasound screen
Arterial cannulation time | During radial artery cannulation (up to 1 hour)
  From needle puncture, to Arterial waveform
Overall Procedure time | During radial artery cannulation (up to 1 hour)
  From ultrasound probe application, to Arterial waveform
Overall success rate | During radial artery cannulation (up to 1 hour)
  Success within 2 skin puncture and within 10 minutes at the chosen radial artery
Malfunction of radial artery catheter | After radial artery cannulation assessed during anesthesia (up to 24 hour)
  Malfunction of Invasive blood pressure monitoring, Sampling
Complication rate | After radial artery cannulation assessed up to PACU, PICU stay (up to 24 hour)
  Hematoma, Distal ischemia, Spasm accessed by ultrasound
Operator's experience | During radial artery cannulation (up to 1 hour)
  The prior experience of the operator's in ultrasound-guided vascular cannulation (5-10 cannulations, 10-30 cannulations, 30-50 cannulations, 50-100 cannulations)
Operator's satisfaction | During radial artery cannulation (up to 1 hour)
  Operator's satisfaction, 5 scale (Worst, Poor, Acceptable, Good, Best)

CONTACTS AND LOCATIONS:
Overall Officials: Jin-Tae Kim, MD, PhD, Principal Investigator — Seoul National University Hospital
Locations (1):
- Jin-Tae Kim, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] White L, Halpin A, Turner M, Wallace L. Ultrasound-guided radial artery cannulation in adult and paediatric populations: a systematic review and meta-analysis. Br J Anaesth. 2016 May;116(5):610-7. doi: 10.1093/bja/aew097. PMID 27106964
- [Background] Kim EH, Lee JH, Song IK, Kim JT, Lee WJ, Kim HS. Posterior Tibial Artery as an Alternative to the Radial Artery for Arterial Cannulation Site in Small Children: A Randomized Controlled Study. Anesthesiology. 2017 Sep;127(3):423-431. doi: 10.1097/ALN.0000000000001774. PMID 28682811
- [Background] Cuper NJ, de Graaff JC, Hartman BJ, Verdaasdonk RM, Kalkman CJ. Difficult arterial cannulation in children: is a near-infrared vascular imaging system the answer? Br J Anaesth. 2012 Sep;109(3):420-6. doi: 10.1093/bja/aes193. Epub 2012 Jun 26. PMID 22735300
- [Background] Ishii S, Shime N, Shibasaki M, Sawa T. Ultrasound-guided radial artery catheterization in infants and small children. Pediatr Crit Care Med. 2013 Jun;14(5):471-3. doi: 10.1097/PCC.0b013e31828a8657. PMID 23628835
- [Background] Song IK, Choi JY, Lee JH, Kim EH, Kim HJ, Kim HS, Kim JT. Short-axis/out-of-plane or long-axis/in-plane ultrasound-guided arterial cannulation in children: A randomised controlled trial. Eur J Anaesthesiol. 2016 Jul;33(7):522-7. doi: 10.1097/EJA.0000000000000453. PMID 26986774
- [Background] Maruyama K, Watanabe E, Kin T, Saito K, Kumakiri A, Noguchi A, Nagane M, Shiokawa Y. Smart Glasses for Neurosurgical Navigation by Augmented Reality. Oper Neurosurg. 2018 Nov 1;15(5):551-556. doi: 10.1093/ons/opx279. PMID 29373710
- [Background] Ueda K, Puangsuvan S, Hove MA, Bayman EO. Ultrasound visual image-guided vs Doppler auditory-assisted radial artery cannulation in infants and small children by non-expert anaesthesiologists: a randomized prospective study. Br J Anaesth. 2013 Feb;110(2):281-6. doi: 10.1093/bja/aes383. Epub 2012 Nov 14. PMID 23151422
- [Background] Anantasit N, Cheeptinnakorntaworn P, Khositseth A, Lertbunrian R, Chantra M. Ultrasound Versus Traditional Palpation to Guide Radial Artery Cannulation in Critically Ill Children: A Randomized Trial. J Ultrasound Med. 2017 Dec;36(12):2495-2501. doi: 10.1002/jum.14291. Epub 2017 Jul 8. PMID 28688136
- [Derived] Kim JT, Park JB, Kang P, Ji SH, Kim EH, Lee JH, Kim HS, Jang YE. Effectiveness of head-mounted ultrasound display for radial arterial catheterisation in paediatric patients by anaesthesiology trainees: A randomised clinical trial. Eur J Anaesthesiol. 2024 Jul 1;41(7):522-529. doi: 10.1097/EJA.0000000000001985. Epub 2024 Mar 21. PMID 38517311